CLINICAL TRIAL: NCT01619618
Title: Evaluation of Polymorphisms and Mutations in Genes Postulated to Alter the Efficacy of Gefitinib in Samples From E1302
Brief Title: Studying Biomarkers in Samples From Patients With Recurrent or Metastatic Head and Neck Cancer Treated on E1302 Trial
Status: Completed | Type: Observational
Sponsor: Eastern Cooperative Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CDR0000734898; ECOG-E1302T1
Record Dates: First submitted 2012-06-12; First posted 2012-06-14 (Estimated); Last update posted 2017-05-17 (Actual); Status verified 2017-05

CONDITIONS: Head and Neck Cancer
Keywords: recurrent squamous cell carcinoma of the hypopharynx; stage IV squamous cell carcinoma of the hypopharynx; recurrent squamous cell carcinoma of the larynx; stage IVA squamous cell carcinoma of the larynx; stage IVB squamous cell carcinoma of the larynx; stage IVC squamous cell carcinoma of the larynx; recurrent squamous cell carcinoma of the lip and oral cavity; stage IVA squamous cell carcinoma of the lip and oral cavity; stage IVB squamous cell carcinoma of the lip and oral cavity; stage IVC squamous cell carcinoma of the lip and oral cavity; recurrent metastatic squamous neck cancer with occult primary; recurrent squamous cell carcinoma of the nasopharynx; stage IV squamous cell carcinoma of the nasopharynx; recurrent squamous cell carcinoma of the oropharynx; stage IVA squamous cell carcinoma of the oropharynx; stage IVB squamous cell carcinoma of the oropharynx; stage IVC squamous cell carcinoma of the oropharynx; recurrent squamous cell carcinoma of the paranasal sinus and nasal cavity; stage IVA squamous cell carcinoma of the paranasal sinus and nasal cavity; stage IVB squamous cell carcinoma of the paranasal sinus and nasal cavity; stage IVC squamous cell carcinoma of the paranasal sinus and nasal cavity; recurrent salivary gland cancer; stage IVA salivary gland cancer; stage IVB salivary gland cancer; stage IVC salivary gland cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck; Salivary Gland Neoplasms | interventions — Polymerase Chain Reaction; Amplified Fragment Length Polymorphism Analysis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other

INTERVENTIONS:
Genetic: mutation analysis
Genetic: polymerase chain reaction
Genetic: polymorphism analysis
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Studying samples of blood and tissue from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer. It may also help doctors predict how patients will respond to treatment.

PURPOSE: This laboratory study is looking at biomarkers in samples from patients with recurrent or metastatic head and neck cancer treated on ECOG-E1302 trial.

DETAILED DESCRIPTION:
OBJECTIVES:

* To evaluate the frequency of ATP-binding cassette, sub-family G (WHITE), member 2 (ABCG2), met proto-oncogene (hepatocyte growth factor receptor) (c-MET), and v-Ki-ras2 Kirsten rat sarcoma viral oncogene homolog (K-ras) polymorphisms or mutations in this study population and the predictiveness of these polymorphisms on survival, time to progression, response rate, and toxicities.

OUTLINE: Archived tumor tissue and peripheral blood mononuclear cells are analyzed for the frequency of ABCG2, c-MET, and K-ras polymorphisms or mutations by polymerase chain reaction (PCR). Results are then correlated with patients' clinical outcomes and toxicity.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Patients diagnosed with recurrent or metastatic head and neck cancer treated on Eastern Cooperative Oncology Group (ECOG)-E1302 trial

  * Patients treated with docetaxel with versus without gefitinib
* Existing paraffin blocks and peripheral blood mononuclear cells

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Samples from patients accrued to E1302 from which specimens were submitted for research.
Sampling Method: Non-Probability Sample
Enrollment: 183 (Actual)
Dates: Start 2012-06-01 (Actual); Primary Completion 2012-07-01 (Actual); Study Completion 2012-07-01 (Actual)

PRIMARY OUTCOMES:
The prevalence of c-MET, ABCG2, and K-ras polymorphisms or mutation status summarized by frequency and percentage for all samples | 1 year
Association of c-MET, ABCG2, and K-ras polymorphisms or mutation status with toxicity using Fisher's exact test | 1 year
Association between biomarkers and time to event distribution estimated by by Kaplan-Meier and estimated by log-rank tests | 1 year
Association between biomarkers and clinical endpoints using logistic regression model and Cox proportional hazards | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Jill Kolesar, PharmD, Principal Investigator — University of Wisconsin, Madison